CLINICAL TRIAL: NCT03446937
Title: Effect of Antenatal Corticosteroids on Neonatal Morbidity.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahmadu Bello University Teaching Hospital (Other)
Responsible Party: Principal Investigator, Anisah Yahya, Lecturer I/Fellow, Ahmadu Bello University Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: AhmaduBUTH
Record Dates: First submitted 2018-02-05; First posted 2018-02-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-12

CONDITIONS: Neonatal Respiratory Distress Syndrome
Keywords: Antenal corticosteroids; Late preterm delivery; Neonatal morbidity
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn | interventions — dexamethasone 21-phosphate; betamethasone sodium phosphate; Dosage Forms; Water; Injections

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexamethasone sodium phosphate injection (Experimental): Intervention: Drug: Dexamethasone sodium phosphate injection Two doses Intramuscular Dexamethasone sodium phosphate 12mg given12 hours apart. (produced by Taizhou Overseas International Ltd. 126-128 Qingnian Road Jiaojiang, Taizhou, Zhejiang, China)
  Interventions: Drug: Dexamethasone Sodium Phosphate Injection
- Betamethasone sodium phosphate injection (Experimental): Intervention: Drug: Betamethasone sodium phosphate injection Two doses of intramuscular betamethasone sodium phosphate 12mg given 12 hours apart. (obtained from Twinbrook pkwy, Rockville, MD Singapore. CAT No 1068004, Lot: R004e0)
  Interventions: Drug: Betamethasone Sodium Phosphate Injection (Medication)
- Water for injection (Placebo Comparator): Intervention. Drug: Water for injection. Two doses of intramuscular water for injection given 12 hours apart.
  Interventions: Drug: Water for injection

INTERVENTIONS:
Drug: Dexamethasone Sodium Phosphate Injection — Dexamethasone sodium phosphate injection 12 mg X doses to be given 12 hours apart
  Other Names: Pemadex
  Arms: Dexamethasone sodium phosphate injection
Drug: Betamethasone Sodium Phosphate Injection (Medication) — betamethasone sodium phosphate injection12mg X 2 doses given 12 hours apart
  Arms: Betamethasone sodium phosphate injection
Drug: Water for injection — Two doses of intramuscular injection of water for injection given 12 hours apart
  Other Names: Juhel water for injection
  Arms: Water for injection

SUMMARY:
It will be a randomized controlled trial. There will be two study groups. Study group 1 will be given dexamethasone while study group 2 will be given betamethasone. The control group will be given placebo.

DETAILED DESCRIPTION:
The study will be a double blind randomised controlled trial. There will be two study groups and one control group.

The first study group will be the pregnant women at risk of late preterm birth that will receive antenatal corticosteroids in the form of intramuscular dexamethasone sodium phosphate.

The second study group will be the pregnant women at risk of late preterm birth that will receive antenatal corticosteroids in the form of intramuscular betamethasone sodium phosphate.

The control group will be pregnant women at risk of late preterm birth that will be given intramuscular water for injection.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women at 34 weeks 0 days to 36 weeks 6 days of gestation and a probability of delivery in the late preterm period irrespective of diagnosis who give consent.
* Pregnant women at 34 weeks 0 days to 36 weeks 6 days of gestation scheduled for elective/emergency delivery in the late preterm period irrespective of indication and route of delivery who give consent.

Exclusion Criteria:

* Evidence of Chrioamnionitis.
* Evidence of foetal distress.
* History of use of antenatal corticosteroids in index pregnancy.
* Women who do not give consent.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Neonatal Respiratory distress syndrome | Within the first 72 hours of life
  Tachypnoea with grunting, recession, or nasal flaring with diffuse reticulogranular infiltrate on X-ray and oxygen requirement.

SECONDARY OUTCOMES:
Transient tachypnoea of the newborn: | Within the first 72 hours after delivery/birth
  As determined by local treatment protocols at Ahmadu Bello University Teaching Hospital
Admission into neonatal intensive care unit. | Within the first 72 hours after delivery/birth
  As determined by local treatment protocols at Ahmadu Bello University Teaching Hospital
2. Admission into neonatal intensive care unit. Apnoea. | Within the first 72 hours after delivery/birth
  As determined by local treatment protocols at Ahmadu Bello University Teaching Hospital

CONTACTS AND LOCATIONS:
Overall Officials: Anisah Yahya, MBBS, Principal Investigator — Ahmadu Bello University
Locations (1):
- Ahmadu Bello University Teaching Hospital Shika-Zaria, Zaria, Kaduna State, Nigeria

IPD SHARING:
Plan to Share IPD: Yes
The outcome will be shared
Supporting Information: Study Protocol, CSR
Time Frame: Data will be made available 6 months after completion and will be made available for 6 months
Access Criteria: It will be shared on request

REFERENCES:
- [Derived] Yahya A, Sulayman HU, Abdulkadir I, Lawal BB. Effect of Antenatal Corticosteroids in Late Preterm Delivery on Neonatal Respiratory Morbidity: A Randomized Controlled Trial. Niger Med J. 2023 Oct 21;64(4):532-544. doi: 10.60787/NMJ-64-4-297. eCollection 2023 Jul-Aug. PMID 38952884